CLINICAL TRIAL: NCT07038278
Title: 5-AminoLevulinic Acid Aided Resection Margins in Sarcoma (5-ALARMS)
Brief Title: 5-AminoLevulinic Acid Aided Resection Margins in Sarcoma
Acronym: 5-ALARMS
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: NX Development Corp (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 24-2149.cc
Record Dates: First submitted 2025-04-09; First posted 2025-06-26 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Soft Tissue Sarcoma (STS)
Keywords: soft tissue sarcoma; fluorescence
MeSH Terms: conditions — Sarcoma | interventions — Aminolevulinic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention Group (Experimental): Patients diagnosed with Federation Nationale des Centres de Lutte Contre le Cancer (FNCLCC) Grade 2 or 3 soft tissue sarcomas who undergo surgical resection will be administered 20 mg/kg body weight of 5-ALA orally at 3-4 hours prior to anesthesia.
  Interventions: Drug: 5-ALA

INTERVENTIONS:
Drug: 5-ALA — 5-ALA), also known by its brand name Gleolan, is an intermediate in the heme synthesis pathway that has been studied in tumor resections, especially in intracranial tumor resections. One advantage of intraoperative visualization with 5-ALA is the ability to directly visualize fluorescent tumor in the surgical field using a headset-mounted devices with fluorescence in the visual wavelength in real-time.
  Other Names: Gleolan

SUMMARY:
The goal of this study is to learn if the intervention using a fluorescent agent 5-Aminolevulinic acid (5-ALA) to aid in the surgical approach to visualize the soft-tissue sarcoma (STS) during surgical resection. 5-ALA goes through the blood stream and into the tumor tissue allowing it to light up when the surgeon uses a special light in the operating room. The technique is called 5-ALA fluorescence-guided surgery (FGS). The main question aims to answer if 5-ALA provide intraoperative fluorescent visualization of soft-tissue sarcoma versus surrounding tissue and demonstrate the efficacy of tumor and surgical margin resections by a gross and histological analysis of fluorescing and non-fluorescing samples immediately after removal. Participants will be asked to orally administer 5-ALA three to four hours prior to surgery in preoperative area.

ELIGIBILITY:
Inclusion Criteria:

1. Histological confirmation of any subtype of primary Grades 2 or 3 soft tissue sarcomas (STS), per biopsy evaluation by a pathologist, according to Fédération Nationale des Centres de Lutte Contre le Cancer (FNCLCC).
2. Treatment decision includes planned surgical resection of STS.
3. Age ≥18 years at time of consent.
4. ECOG Performance Status 0 - 1.
5. Hematology and blood chemistry parameters defined by:

   1. Leukocytes ≥ 3 × 10(9)/L
   2. Absolute neutrophil count ≥ 1.5 × 10(9)/L
   3. Platelets ≥ 100 × 109/L, transfusions may be used to raise platelets to ≥ 100 × 10(9)/L (no washout required)
   4. Hemoglobin ≥ 9 g/dL, transfusions may be used to raise Hgb to ≥ 9 g/dL (no washout required)
   5. Total bilirubin ≤ 1.5 × institutional upper limit of normal (ULN)
   6. Aspartate transaminase (AST) / alanine transaminase (ALT) ≤ 2.5 × institutional ULN
   7. Creatinine within normal institutional limits OR creatinine clearance ≥ 30 mL/min/1.73 m2 for patients with creatinine above institutional ULN
6. Participants of reproductive potential must agree to using adequate contraception (e.g., hormonal or barrier method of birth control; abstinence, an intrauterine device) for the duration of study participation (including dosing interruptions) and up to 42 days after end of study intervention; or be surgically sterilized (e.g., hysterectomy, tubal ligation, or vasectomy).
7. Ability to swallow study agent.
8. Ability to understand and willingness to sign an informed consent form.
9. Ability and stated willingness to adhere to the study visit schedule and other protocol procedures/requirements for the duration of the study.

Inclusion of Minorities and Other Underrepresented Populations Recruitment is open and encouraged to all genders, all minorities, and underrepresented populations. Although distributions may vary by disease type, our recruitment procedures have been developed to enroll participants who are representative of the respective target population.

Exclusion Criteria:

1. Acute/chronic forms of porphyria.
2. Uncontrolled, known concurrent illness, including but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness.
3. Patient has had chemotherapy, tumor resection, or radiation treatment ≤ 21 days prior to surgery.
4. Simultaneous participation in another clinical trial ≤ 21 days of enrollment or during the duration of the study period.
5. Planned use of other potentially phototoxic substances (e.g., St. John's wort, griseofulvin, thiazide diuretics, sulfonylureas, phenothiazines, sulfonamides, quinolones and tetracyclines), and topical preparations containing aminolevulinic acid (5-ALA) for 24 hours during the perioperative period (defined as 24 hours prior to surgery to up to 24 hours post-surgery).
6. Pregnant or planning to become pregnant during study participation or breastfeeding.
7. Any condition that is in the opinion of the investigator would prohibit the understanding or rendering of informed consent or interfere with the participant's safety or compliance while on trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Demonstrate the feasibility of 5-ALA aided fluorescent visualization of soft tissue sarcomas versus surrounding tissues | From enrollment to 2 weeks
  Patients will receive 5-ALA administered in the preoperative area. Surgical resection of the soft tissue sarcoma will be done as per standard of care.
  A fluorescent headset will be turned on at defined time points below and tumor fluorescence will be noted (yes or no):
  1. prior to skin incision
  2. once dissection has reached fascial layer
  3. when 50% of the tumor superficial-to-deep has been dissected
  4. following complete resection of the tumor.
Surgeon survey results of intraoperative tumor fluorescence | perioperative/periprocedural
  Surgeons will fill out survey (yes or no) to answer following intraoperative assessment questions:
  1. if the tumor demonstrated fluorescence from 5-ALA
  2. Was the tumor fluorescence discernable from normal tissue.
  3. Did the 5-ALA use increase or decrease the resection amount
  4. Was the equipment was easy to use

SECONDARY OUTCOMES:
Demonstrate the efficacy of 5-ALA fluorescence in tumor resections by a histological analysis of non-fluorescing samples after tumor removal | Day of Surgery
  The sarcoma tumor will then be hemisected immediately after resection in pathology lab.
  The fluorescent headset will be used to identify areas of fluorescence in the tumor.
  Multiple samples (3mm punch) will be taken from nonfluorescent areas and placed on slides:
  Histologic analysis will evaluate for viable tumor cells (%). For this, Sensitivity will be considered as the proportion of cells who had viable tumor that fluoresced, with specificity as the proportion of cells that had non-viable tumor without fluorescence.
Demonstrate the efficacy of 5-ALA fluorescence in tumor resections by a histological analysis of fluorescing samples after tumor removal | Day of surgery
  Description: The sarcoma tumor will then be hemisected immediately after resection in pathology lab. The fluorescent headset will be used to identify areas of fluorescence in the tumor. Multiple samples (3mm punch) will be taken from these fluorescent areas in the tumor and placed on slides: Specific to the margins and include the relevant presence of fluorescence (yes/no), cancer cells(%). For this, Sensitivity will be considered as the proportion of cancerous cells that fluoresced, with specificity as the proportion of non-cancerous cells that did not.
Demonstrate the efficacy of 5-ALA fluorescence in tumor resections by a histological analysis of fluorescing samples after tumor removal | Day of surgery
  The sarcoma tumor will then be hemisected immediately after resection in pathology lab.
  The fluorescent headset will be used to identify areas of fluorescence in the tumor.
  Multiple samples (3mm punch) will be taken from these fluorescent areas in the tumor and placed on slides:
  These will be specific to the tumor and include the relevant presence of fluorescence (yes/no), viable tumor cells (%). For this, Sensitivity will be considered as the proportion of cells who had viable tumor that fluoresced, with specificity as the proportion of cells that had non-viable tumor without fluorescence.
Determine oncologic outcomes for patients enrolled | From enrollment to 2 years
  Local recurrence free survival will be determined from time of surgery and with use of MRI with contrast
Patient Reported Outcomes | From enrollment to 2 years
  Patient Reported Outcomes Measurement Information System (PROMIS) patient reported outcome measure.
Patient Reported Outcomes | From enrollment to 2 years.
  Toronto Extremity Salvage Score (TESS) patient reported outcome measure.
Patient Reported Outcomes | From enrollment to 2 years.
  Visual Analog Scales (VAS) patient reported outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Thorpe, MD, FACS, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Teixidor P, Arraez MA, Villalba G, Garcia R, Tardaguila M, Gonzalez JJ, Rimbau J, Vidal X, Montane E. Safety and Efficacy of 5-Aminolevulinic Acid for High Grade Glioma in Usual Clinical Practice: A Prospective Cohort Study. PLoS One. 2016 Feb 17;11(2):e0149244. doi: 10.1371/journal.pone.0149244. eCollection 2016. PMID 26885645
- [Background] Giantini-Larsen AM, Kharas N, Pisapia D, Schwartz TH. Histology of high-grade glioma samples resected using 5-ALA fluorescent headlight and loupe combination. Acta Neurochir (Wien). 2023 Feb;165(2):567-575. doi: 10.1007/s00701-023-05496-8. Epub 2023 Jan 19. PMID 36656388
- [Background] Stummer W, Pichlmeier U, Meinel T, Wiestler OD, Zanella F, Reulen HJ; ALA-Glioma Study Group. Fluorescence-guided surgery with 5-aminolevulinic acid for resection of malignant glioma: a randomised controlled multicentre phase III trial. Lancet Oncol. 2006 May;7(5):392-401. doi: 10.1016/S1470-2045(06)70665-9. PMID 16648043
- [Background] Schupper AJ, Baron RB, Cheung W, Rodriguez J, Kalkanis SN, Chohan MO, Andersen BJ, Chamoun R, Nahed BV, Zacharia BE, Kennedy J, Moulding HD, Zucker L, Chicoine MR, Olson JJ, Jensen RL, Sherman JH, Zhang X, Price G, Fowkes M, Germano IM, Carter BS, Hadjipanayis CG, Yong RL. 5-Aminolevulinic acid for enhanced surgical visualization of high-grade gliomas: a prospective, multicenter study. J Neurosurg. 2021 Oct 8;136(6):1525-1534. doi: 10.3171/2021.5.JNS21310. Print 2022 Jun 1. PMID 34624862
- [Background] Mahmoudi K, Garvey KL, Bouras A, Cramer G, Stepp H, Jesu Raj JG, Bozec D, Busch TM, Hadjipanayis CG. 5-aminolevulinic acid photodynamic therapy for the treatment of high-grade gliomas. J Neurooncol. 2019 Feb;141(3):595-607. doi: 10.1007/s11060-019-03103-4. Epub 2019 Jan 18. PMID 30659522
- [Background] Guder WK, Hartmann W, Buhles C, Burdack M, Busch M, Dunker N, Hardes J, Dirksen U, Bauer S, Streitburger A. 5-ALA-mediated fluorescence of musculoskeletal tumors in a chick chorio-allantoic membrane model: preclinical in vivo qualification analysis as a fluorescence-guided surgery agent in Orthopedic Oncology. J Orthop Surg Res. 2022 Jan 15;17(1):34. doi: 10.1186/s13018-022-02931-x. PMID 35033148
- [Background] Kenan S, Liang H, Goodman HJ, Jacobs AJ, Chan A, Grande DA, Levin AS. 5-Aminolevulinic acid tumor paint and photodynamic therapy for myxofibrosarcoma: an in vitro study. J Orthop Surg Res. 2020 Mar 5;15(1):94. doi: 10.1186/s13018-020-01606-9. PMID 32138774
- [Background] Endo M, Lin PP. Surgical margins in the management of extremity soft tissue sarcoma. Chin Clin Oncol. 2018 Aug;7(4):37. doi: 10.21037/cco.2018.08.10. PMID 30173528